CLINICAL TRIAL: NCT07278752
Title: Social Media Concerns Related to Emotional Experiences in Naturalistic Settings (SCREENS)
Acronym: SCREENS
Status: Not yet recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Madhukar H. Trivedi, MD, Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU20252066; R21MH142320-01 (NIH)
Record Dates: First submitted 2025-11-19; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Depression in Adolescence; Suicidal Ideation; Social Media Addiction; Mental Health Issue
MeSH Terms: conditions — Suicidal Ideation; Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to advance understanding of the relationships between social media use (SMU) and internalizing symptoms among a diverse sample of depressed and/or suicidal youth. Youth (ages 13-18) enrolled in the TX-YDSRN registry study will be recruited for participation in SCREENS. After reviewing the Information Sheet, participants will complete baseline measures assessing internalizing symptoms (e.g., depression, anxiety, suicidal ideation/behavior), and trauma history. They will then complete ecological momentary assessments (EMAs) twice daily for 30 days via the mHealth app, capturing internalizing symptoms, emotional responses to social media, and in-person social support. The mHealth app will also collect the amount of social media use during this 30-day period. From Month 1 through Month 6, participants will receive monthly self-report surveys administered through REDCap.

100 participants

This study will enroll youth from the TX-YDSRN registry study who meet all the following criteria:

* Be between 13 and 18 years of age at the time of enrollment.
* Be currently enrolled in the TX-YDSRN registry study and willing to allow sharing of data from that study.
* Own a smartphone and agree to download and use the study mHealth application for the duration of study participation.
* Be willing and able to participate in all study requirements and allocate sufficient time to complete study questionnaires and measures.

Visits include a Screening Visit, Baseline Visit, EMA 2x daily for 30 days, 6 remote follow-up survey visits.

Multiple streams of outcome measures will be utilized for this protocol, including self-report measures, research assessor-completed measure, and EMA measures.

Adverse event (AE) recording, 9 item Patient Health Questionnaire Adolescent Version (PHQ-A), Concise Health Risk Tracking Self Report (CHRT-SR).

DETAILED DESCRIPTION:
The study aims to enroll 100 participants recruited from the TX-YDSRN registry study. TX-YDSRN registry study, an ongoing state-wide longitudinal data repository funded by Texas Child Mental Healthcare Consortium (TCMHCC). TX-YDSRN is comprised of 12 participating HRIs across Texas.

Eligible and active TX-YDSRN participants will be invited to participate in this study. Efforts will be made to ensure a diverse and representative sample, including participants of varying sexes, ethnicities, races, and socioeconomic backgrounds. The TX-YDSRN's established recruitment network and community partnerships since 2020 support broad and inclusive enrollment.

Advances in mobile health (mHealth) technologies offer new ways to monitor depression and suicidal ideation outside of clinical settings. Through smartphones and devices from wearable health technology leaders such as Garmin or Fitbit, this study aims to remotely track clinical indicators among youth. These technologies collect data such as physical activity, social interaction, sleep, social media experiences, social media use amount, and mood in real-time, providing an ecologically valid picture of the participants' daily lives. This approach can enhance early detection of clinical deterioration, empowering both participants and caregivers with timely, actionable feedback.

Using HIPAA-compliant software on smartphones, the app will track digital markers such as location, movement, call/text frequency, screen time, and survey responses as proxies for social interaction, in-person social support, anxiety, suicidal ideation/behavior, emotional responses to social media, and mood. Data is encrypted, stored on secure servers ensuring confidentiality. Similarly, wearables will track digital biomarkers such as sleep patterns, heart rate, and activity levels. Together, these metrics offer continuous, longitudinal data on various potential markers for physical and psychological health such as the following:

* Activity Levels: Reduced physical activity and social engagement may indicate worsening depression. Tracking changes in the radius of daily movement can help detect reduced interest and motivation to engage in important or valued activities.
* Sleep Patterns: Sleep issues (insomnia, hypersomnia, disruption, restlessness) often signal mood changes. By monitoring sleep latency, duration, and quality, we can identify early warning signs of depression.
* Social Interaction: Decreases in communication frequency and network size, changes in screen time, can indicate social withdrawal.
* Mood Variability: Regular assessments of mood, fatigue, and energy help capture emotional variability. Non-responsiveness itself can be a potential marker of worsening of depression.

Social media use amount is passive data that will be collected through mHealth. mHealth will also automatically track duration of app use (seconds) by type of platform and will tell us actual usage (on screen) rather than those running in the background. mHealth will constantly collect data is the app is open and running in the background of the subject's device. These data will be collected constantly for the 1-month period during which Ecological Momentary Assessment Measures (EMA) data are also collected on social media experiences.

Given the study's integration of mobile device monitoring, several strategies will be implemented to enhance participant engagement and retention throughout study participation:

* Mobile Notifications: Participants will receive Ecological Momentary Assessment (EMA) prompts via their mobile devices multiple times per day. These notifications will remind participants to complete assigned tasks, with automated follow-up reminders to encourage timely completion.
* Follow-Up for Non-Response: Participants who do not respond to EMA prompts for more than 48 hours will be contacted by research staff via phone, text message, or email. those proactive check ins will aim to re-engage participants, identify potential barriers, and trouble shoot any technical issues (e.g., adjusting notification settings, reinstallation of the app, or supporting participants who have transitioned to a new device).
* Incentive Structure: A structured incentive plan will be employed to promote consistent engagement and adherence. Participants will be eligible for incremental compensation tied to EMA completion rates, with additional bonus payments provided for high completion percentages across the study period.

Regular communication will be maintained through a combination of phone calls, emails, text messages, and mailed reminders.

Duration of Participation and Visit Schedule Enrollment of 100 subjects is expected to take place over approximately 1 year. Enrolled participants will be involved in the study for 6 months. Visits include a Screening Visit, Baseline Visit, EMA (2 times per day for 30 days), 6 monthly remote follow-up visits.

Outcome Measures Multiple streams of outcome measures will be utilized for this protocol, including self-reported, assessor-completed measures and EMA.

Ecological Momentary Assessment Measures:

The EMA survey administered through the mHealth application will include validated EMA items for Social Media factors of Social Media experiences (positive and negative ERSM) and for social context (adapted from an EMA measure of positive and negative in-person interactions). Primary outcomes will be collected twice daily, morning and evening, and will include items assessing mood and anxiety as well as the 3-item suicidal thoughts subscale of the CHRT-SR16. Participants will answer 5 questions morning and evening related to depression, anxiety, and suicidal ideation. For depression, youth will select which emoticon best represents their current mood (e.g., smiley face, neutral face, frowny face). For anxiety, the question is item 1 from GAD-7. The suicidal ideation questions are items 14-16 on the CHRT-SR16.

Emotional Responses to Social Media (ERSM):

Emotional experiences related to online experiences will be assessed using the Emotional Responses to Social Media (ERSM) scale, which assesses both positive (e.g., "How much did you feel happy or excited because of a positive interaction?") and negative (e.g., "How much did you feel sad or hurt because of a negative interaction?") experiences with social media use. ERSM items include those used in our consultant's prior research and developed based on the ERSM. Four of these items focus on dyadic positive and negative online social interactions. Three items focus on more general social impression. We will explore these separate social media experience constructs to get a more nuanced understanding of types of social media experiences. ERSM questions will only be included in the evening survey.

Questions related to in-person social experiences Items assessing positive and negative in-person interactions will ask participants to think about the most influential offline social interaction they had and rate it as either positive, negative, or mixed. Participants also have the option if they did not have an in-person interaction that day. Based on their response, participants will receive additional questions asking what made the interaction positive or negative and to rate the experience on a scale from 0-10. Questions regarding in-person interactions will only be included in the evening survey.

Further context concerning in-person social experiences will be derived from the Traumatic Events Screening Inventory for Children (TESI-C) clinical interview, which provides information on victimization experiences.

ELIGIBILITY:
Inclusion Criteria:

1. Be between 13 and 18 years of age at the time of enrollment.
2. Be currently enrolled in the TX-YDSRN registry study and willing to allow sharing of data from that study.
3. Own a smartphone and agree to download and use the study mHealth application for the duration of study participation.
4. Be willing and able to participate in all study requirements and allocate sufficient time to complete study questionnaires and measures.

Exclusion Criteria:

1. Have medical, psychiatric, or other condition for which study participation would not be in their best interest or that could interfere or confound study assessments.
2. Require immediate psychiatric hospitalization or present an imminent suicide risk at the time of screening.
3. Unwilling or unable to download or comply with mHealth app requirements.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will leverage the existing Texas Youth Depression and Suicide Research Network (TX-YDSRN) Participant Registry NCT04572321, a natural-history longitudinal data repository of youth with depression and/or suicidal ideation or behavior across 12 Health Related Institutions (HRIs) in Texas. 100 hundred participants aged 13 to 18 years old will be recruited and enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Concise Health Risk Tracking Self-Report (CHRT-SR) | 6 months
  The CHRT is a scale that evaluates specific thoughts about suicide and thoughts and feelings associated with an increased risk for suicide. The self-report CHRT is a 16-item scale that evaluates specific thoughts about suicide and thoughts and feelings associated with an increased risk for suicide. Its psychometric properties have been well-established in children and adolescents.
Patient Health Questionnaire-A (PHQ-A) | 6 months
  The PHQ-A is a nine-item, self-report inventory that assesses for symptoms in all nine symptom domains of a major depressive episode. It is the PHQ-9 modified for adolescents 12-18 years
Generalized Anxiety Disorder Scale - 7 items (GAD-7) | 6 months
  The GAD-7 is self-report that assesses for symptoms in 7 symptom domains of generalized anxiety, with an additional question on anxiety-related functional impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar Trivedi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No